CLINICAL TRIAL: NCT06233526
Title: Individualized Treatment of Pediatric Relasped and Refractory Acute Myeloid Leukemia Based on Transcriptomic Profile and in Vitro Drug Sensitivity Test
Brief Title: Individualized Treatment of Pediatric R/R AML Based on Transcriptomic Profile and in Vitro Drug Sensitivity Test
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: College of Pharmaceutical Science at Zhejiang University (Unknown)
Responsible Party: Principal Investigator, Xiaojun Xu, chief physician, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-IRB-0315-P-01
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Acute Myeloid Leukemia in Children
Keywords: Acute myeloid leukemia; relapsed/refractory; transcriptomic sequencing; drug sensitivity test
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized treatment group (Experimental): Treating the R/R AML patients based on the transcriptomic profile and in vitro drug sensitivity Test
  Interventions: Other: Chemotherapy regiments based on the transcriptomic profile and in vitro drug sensitivity test

INTERVENTIONS:
Other: Chemotherapy regiments based on the transcriptomic profile and in vitro drug sensitivity test — 1. Leukemia cells from newly diagnosed and relapsed children with AML were tested for high throughput in vitro drug sensitivity and resistance.
  2. Combined with multi-omics sequencing technology such as whole exome and transcriptome, the data of drug sensitivity, drug resistance and genomic characteristics of children AML patients were integrated, and the internal rules between drug sensitivity or drug resistance and molecular characteristics such as gene fusion, gene mutation and abnormal gene expression of children AML patients were deeply analyzed, and the molecular characteristics of drug sensitivity in children AML were mapped

SUMMARY:
Acute myeloid leukemia (AML) accounts for about 15% to 20% of childhood leukemia, but the death rate accounts for about 50%. About 20-30% of children with AML did not achieve complete response (CR) after 2 induction treatments, and about 30% of children with CR had relapse within 3 years (including recurrence after hematopoietic stem cell transplantation).Relapsed/refractory (R/R) AML is a major cause of treatment failure and refractory survival. Reinduction chemotherapy for R/R-AML to obtain CR again, followed by hematopoietic stem cell transplantation, is the current treatment. At present, there is no recognized reinduction protocol, and the reinduction remission rate of R/R-AML varies greatly among different treatment regimens, ranging from 23 to 81%. Current guidelines recommend a new combination chemotherapy regimen consisting of new drugs without cross-resistance. This method selects sensitive chemotherapeutic drugs, and then forms a new combination chemotherapy regimen according to the characteristics of drugs, which is the choice of R/R-AML reinduction therapy.This study intends to conduct a clinical study on the individualized treatment of R/R AML patients through in vitro drug sensitivity test combined with patient transcriptomic characteristics.

ELIGIBILITY:
Inclusion Criteria:

- (1) Refractory recurrent acute myeloid leukemia (AML), and after second-line reinduction therapy, such as C+HAG did not reach complete CR.Criteria for complete response, refractory, and recurrence are as follows.

(2) <18 years old; (3) The child had good organ function, could tolerate chemotherapy, and had a physical strength score of 0-3 (WHO standard); (4) Understand the research procedures and voluntarily sign written informed consent.

Exclusion Criteria:

- (1) Acute promyelocytic leukemia, chronic myelogenous leukemia, acute mixed cell leukemia or known central nervous system leukemia; (2) AML associated with congenital syndromes such as Down syndrome, Fanconi anemia, Bloom syndrome, Cole's syndrome, or congenital aplastic anemia; (3) secondary to immunodeficiency or positive for human immunodeficiency virus (HIV); (4) Cardiac and renal function were obviously abnormal, and left ventricular ejection fraction was <50%.

(5) There is active systemic infection; (6) any medical history or concomitant condition that the investigator believes would impair the subject's safe completion of the study; (7) The investigator considers that the subject is medically unfit to receive the investigational drug or is unfit for any other reason; (8) a known or suspected allergy to the subject drug or to any drug administered in connection with this test;

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | 4 weeks
  Complete remission rate after the course of individualized treatment
Event free survival | one year, five years
  The patient's event free survival at one and five years after treatment

SECONDARY OUTCOMES:
Overall Survival | one year, five years
  The patient's overall survival at one and five years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Xu, MD, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Newell LF, Cook RJ. Advances in acute myeloid leukemia. BMJ. 2021 Oct 6;375:n2026. doi: 10.1136/bmj.n2026. PMID 34615640
- [Background] Kim H. Treatments for children and adolescents with AML. Blood Res. 2020 Jul 31;55(S1):S5-S13. doi: 10.5045/br.2020.S002. PMID 32719170
- [Background] Zarnegar-Lumley S, Caldwell KJ, Rubnitz JE. Relapsed acute myeloid leukemia in children and adolescents: current treatment options and future strategies. Leukemia. 2022 Aug;36(8):1951-1960. doi: 10.1038/s41375-022-01619-9. Epub 2022 Jun 6. PMID 35668109
- [Background] Leukemia & Lymphoma Group, Chinese Society of Hematology, Chinese Medical Association. [Chinese guidelines for the diagnosis and treatment of relapsed/refractory acute myelogenous leukemia (2021)]. Zhonghua Xue Ye Xue Za Zhi. 2021 Aug 14;42(8):624-627. doi: 10.3760/cma.j.issn.0253-2727.2021.08.002. No abstract available. Chinese. PMID 34547866
- [Background] Kamens JL, Nance S, Koss C, Xu B, Cotton A, Lam JW, Garfinkle EAR, Nallagatla P, Smith AMR, Mitchell S, Ma J, Currier D, Wright WC, Kavdia K, Pagala VR, Kim W, Wallace LM, Cho JH, Fan Y, Seth A, Twarog N, Choi JK, Obeng EA, Hatley ME, Metzger ML, Inaba H, Jeha S, Rubnitz JE, Peng J, Chen T, Shelat AA, Guy RK, Gruber TA. Proteasome inhibition targets the KMT2A transcriptional complex in acute lymphoblastic leukemia. Nat Commun. 2023 Feb 13;14(1):809. doi: 10.1038/s41467-023-36370-x. PMID 36781850
- [Result] Du W, Xia Z, Luo Z, Chen Y, Bing S, Wang W, Zhang X, Zhou Z, Zhang J, Cao J, Yang B, He Q, Shao X, Xu X, Ying M. A novel gene fusion RUNX1/ZNF423 promotes leukemic relapse of NUP98-rearranged AML. Leukemia. 2023 Nov;37(11):2286-2291. doi: 10.1038/s41375-023-02024-6. Epub 2023 Sep 15. No abstract available. PMID 37714925